CLINICAL TRIAL: NCT03938246
Title: A Phase 2, Multi-Center, Single-Blind, Randomized, Placebo-Controlled Study of TVB-2640 in Subjects With Non-Alcoholic Steatohepatitis (FASCINATE-1)
Brief Title: Study of TVB-2640 in Subjects With Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3V2640-CLIN-005
Record Dates: First submitted 2019-04-24; First posted 2019-05-06 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: MASLD/MASH (Metabolic Dysfunction-Associated Steatotic Liver Disease / Metabolic Dysfunction-Associated Steatohepatitis)
Keywords: NASH; Non-Alcoholic Steatohepatitis; Fatty Liver Disease; Fatty Liver; Liver Diseases; FASN; Fatty Acid Synthase Inhibitor
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Diseases | interventions — TVB-2640

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to experimental or placebo arms.
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- TVB-2640 25 mg (US) (Experimental): Subjects randomly assigned to receive the study drug will take TVB-2640 tablet orally every day for 12 week treatment period. The dose is to be taken at the same time of the day, with each dose separated by 24 hours (±4 hours).
  Interventions: Drug: TVB-2640 25 mg (US)
- TVB-2640 50 mg (US) (Experimental): Subjects randomly assigned to receive the study drug will take TVB-2640 tablet orally every day for 12 week treatment period. The dose is to be taken at the same time of the day, with each dose separated by 24 hours (±4 hours).
  Interventions: Drug: TVB-2640 50 mg (US)
- Placebo (US) (Placebo Comparator): Subjects randomly assigned to placebo will receive placebo tablets orally once a day under the same conditions and frequency as described for TVB-2640.
  Interventions: Drug: Placebo (US)
- TVB-2640 50 mg (China) (Experimental): Subjects randomly assigned to receive the study drug will take TVB-2640 tablet orally every day for 12 week treatment period. The dose is to be taken at the same time of the day, with each dose separated by 24 hours (±4 hours).
  Interventions: Drug: TVB-2640 50 mg (China)
- Placebo (China) (Placebo Comparator): Subjects randomly assigned to placebo will receive placebo tablets orally once a day under the same conditions and frequency as described for TVB-2640.
  Interventions: Drug: Placebo (China)
- TVB-2640 75 mg (US) (Experimental): After completion of Cohorts 1 and 2, and if no stopping criteria are met upon review by the Independent SRC, an additional TVB-2640 75 mg open-label Cohort 3 will open in the US
  Interventions: Drug: TVB-2640 75 mg (US)

INTERVENTIONS:
Drug: TVB-2640 25 mg (US) — Oral dose, tablet, daily dosing
  Arms: TVB-2640 25 mg (US)
Drug: TVB-2640 50 mg (US) — Oral dose, tablet, daily dosing
  Arms: TVB-2640 50 mg (US)
Drug: Placebo (US) — Oral dose, tablet, daily dosing
  Arms: Placebo (US)
Drug: TVB-2640 50 mg (China) — Oral dose, tablet, daily dosing
  Arms: TVB-2640 50 mg (China)
Drug: Placebo (China) — Oral dose, tablet, daily dosing
  Arms: Placebo (China)
Drug: TVB-2640 75 mg (US) — Oral dose, tablet, daily dosing
  Arms: TVB-2640 75 mg (US)

SUMMARY:
This is a Phase 2 multi-center, randomized, single-blind, placebo-controlled study to evaluate the safety and efficacy of TVB-2640 in subjects with non-alcoholic steatohepatitis (NASH), a type of fatty liver disease. Subjects will be randomly assigned to 1 of 2 treatment groups (TVB-2640 at one of three doses or placebo). Following randomization, subjects will begin the 12-week treatment period and will receive once daily TVB-2640 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years with a body mass index (BMI) ≤40 kg/m2.
2. Prior liver biopsy within 24 months of randomization with fibrosis Stage 1 to 3 and a non-alcoholic fatty liver disease (NAFLD) activity score (NAS) of ≥ 4 with at least a score of 1 in each of the following NAS components:

   * Steatosis
   * Ballooning degeneration
   * Lobular inflammation

AND

* Confirmation of ≥ 8% liver fat content on MRI-PDFF.

OR, if prior biopsy is not available:

* Either overweight or obese or diabetic or ALT ≥ 30 U/L or fatty liver on ultrasound and at least one more feature of metabolic syndrome by Adult Treatment Panel III (ATP III) criteria.

AND

* Magnetic resonance elastography (MRE) ≥ 2.5 kPa and MRI-PDFF ≥ 8% during screening.

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for enrollment in the study.

1. History of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening.

   Note: Significant alcohol consumption is defined as average of > 20 g/day in female subjects and > 30 g/day in male subjects.
2. Type 1 diabetes.
3. Uncontrolled Type 2 diabetes defined as:

   * HbA1c ≥ 9.5% during screening. (Subjects with HbA1c ≥ 9.5% may be rescreened).
   * Basal insulin dose adjustment > 10% within 60 days prior to enrollment.
   * Requirement for glucagon-like peptide analogue or a complex oral anti-diabetic (OAD) regimen (3 or more OADs) within 6 months of screening.
   * History of severe hypoglycemia (symptomatic hypoglycemia requiring outside assistance to regain normal neurologic status) within the previous year.

   Note: Individual diabetes regimens will be reviewed by Investigator and may be adjusted based on American Diabetes Association guidelines.
4. Presence of cirrhosis on liver biopsy (Stage 4 fibrosis) or imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2021-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, MD, Principal Investigator — UCSD
Locations (23):
- United States (12):
  - ProSciento, Chula Vista, California
  - Catalina Research Institute, Montclair, California
  - Clinical Trials Research, Sacramento, California
  - University of California San Diego (UCSD), San Diego, California
  - Panax, Miami Lakes, Florida
  - Lucas Research, Morehead City, North Carolina
  - Texas Diabetes and Endocrinology - Austin, Austin, Texas
  - Texas Digestive Disease Consultants - Cedar Park, Cedar Park, Texas
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - Texas Digestive Disease Consultant - Ft Worth, Fort Worth, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - Texas Digestive Disease Consultants - Webster, Webster, Texas
- China (11):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Foshan First People's Hospital, Foshan, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Second Hospital of Nanjing, Nanjing, Jiangsu
  - Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Tongren Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loomba R, Mohseni R, Lucas KJ, Gutierrez JA, Perry RG, Trotter JF, Rahimi RS, Harrison SA, Ajmera V, Wayne JD, O'Farrell M, McCulloch W, Grimmer K, Rinella M, Wai-Sun Wong V, Ratziu V, Gores GJ, Neuschwander-Tetri BA, Kemble G. TVB-2640 (FASN Inhibitor) for the Treatment of Nonalcoholic Steatohepatitis: FASCINATE-1, a Randomized, Placebo-Controlled Phase 2a Trial. Gastroenterology. 2021 Nov;161(5):1475-1486. doi: 10.1053/j.gastro.2021.07.025. Epub 2021 Jul 23. PMID 34310978

RESULTS

PARTICIPANT FLOW:
Groups:
- TVB-2640 25 mg (US); TVB-2640 50 mg (US); TVB-2640 50 mg (China); TVB-2640 75 mg (US): TVB-2640 tablet orally every day for 12 weeks
- Placebo (US); Placebo (China): Placebo tablet orally every day for 12 weeks
Period: Overall Study
Arm/Group | TVB-2640 25 mg (US) | TVB-2640 50 mg (US) | Placebo (US) | TVB-2640 50 mg (China) | Placebo (China) | TVB-2640 75 mg (US)
Started | 33 | 35 | 31 | 21 | 9 | 13
Completed | 27 | 30 | 31 | 20 | 9 | 11
Not Completed | 6 | 5 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The overall number of participants that are provided here are as per safety population.
  Note- The Safety Population consisted of all randomized subjects who received at least 1 dose of study drug. Analysis is based on randomized treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | TVB-2640 25 mg (US) | TVB-2640 50 mg (US) | Placebo (US) | TVB-2640 50 mg (China) | Placebo (China) | TVB-2640 75 mg (US) | Total
Number analyzed (Participants) | 33 | 35 | 31 | 21 | 9 | 13 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 29 | 27 | 19 | 8 | 12 | 122
  >=65 years | 6 | 6 | 4 | 2 | 1 | 1 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 17 | 4 | 3 | 5 | 57
  Male | 18 | 22 | 14 | 17 | 6 | 8 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 24 | 25 | 0 | 0 | 13 | 84
  Not Hispanic or Latino | 11 | 11 | 6 | 21 | 9 | 0 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 35 | 31 | 0 | 0 | 13 | 112
  China | 0 | 0 | 0 | 21 | 9 | 0 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Hepatic Fat Fraction by Magnetic Resonance Imaging Proton Density Fat Fraction (MRI-PDFF) From Baseline
Description: As determined by MRI-PDFF
Time Frame: 12 weeks
Population: Analyses using only subjects in the mITT Population who had data at Baseline and Week 12 for observed relative change values from Baseline to Week 12
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | TVB-2640 25 mg (US) | TVB-2640 50 mg (US) | Placebo (US) | TVB-2640 50 mg (China) | Placebo (China) | TVB-2640 75 mg (US)
Number analyzed (Participants) | 26 | 27 | 23 | 19 | 7 | 7
percent change from baseline | -11.31 (29.837) | -27.59 (28.354) | 2.52 (33.030) | -28.68 (22.265) | -15.63 (30.789) | -35.77 (23.736)

2. Secondary Outcome: Percentage of Subjects With at Least a 30% Reduction in Liver Fat at Week 12.
Description: As determined by MRI-PDFF
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | TVB-2640 25 mg (US) | TVB-2640 50 mg (US) | Placebo (US) | TVB-2640 50 mg (China) | Placebo (China) | TVB-2640 75 mg (US)
Number analyzed (Participants) | 26 | 27 | 23 | 19 | 7 | 7
Participants | 7 | 16 | 3 | 10 | 2 | 4

3. Secondary Outcome: Percentage of Change From Baseline in Alanine Aminotransferase (ALT)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | TVB-2640 25 mg (US) | TVB-2640 50 mg (US) | Placebo (US) | TVB-2640 50 mg (China) | Placebo (China) | TVB-2640 75 mg (US)
Number analyzed (Participants) | 30 | 31 | 29 | 20 | 9 | 7
percentage of change | -2.98 (38.443) | -20.46 (25.935) | 6.82 (37.258) | -28.29 (34.495) | 14.06 (79.621) | -3.296 (42.5397)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The intensity of each AE was assessed by the Investigator according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
Arm/Group | TVB-2640 25 mg (US) | TVB-2640 50 mg (US) | Placebo (US) | TVB-2640 50 mg (China) | Placebo (China) | TVB-2640 75 mg (US)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35 | 0/31 | 0/21 | 0/9 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35 | 0/31 | 0/21 | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 25/33 | 14/35 | 12/31 | 17/21 | 5/9 | 9/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TVB-2640 25 mg (US) (N=33) | TVB-2640 50 mg (US) (N=35) | Placebo (US) (N=31) | TVB-2640 50 mg (China) (N=21) | Placebo (China) (N=9) | TVB-2640 75 mg (US) (N=13)
Headache (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 8 (8) | 2 (2) | 5 (5)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival deposit (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT03938246/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT03938246/SAP_001.pdf